CLINICAL TRIAL: NCT05401331
Title: Effect of Mask Use on Hemodynamic Responses During Exertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Mask and Hemodynamic Responses
Record Dates: First submitted 2022-04-11; First posted 2022-06-02 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Heart Rate; Blood Pressure; Exercise Test; Mask
Keywords: Dyspnea; Mask; Oxygen Saturation; Blood Pressure; Heart Rate; Exercise Test; COVİD-19
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Sphygmomanometers; Masks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodynamic changes due to mask use (Other): Hemodynamic changes due to mask use
  Interventions: Device: Treadmilll; Other: mask
- Hemodynamic responses when we do not use masks (Other): Hemodynamic responses when we do not use masks
  Interventions: Device: Treadmilll

INTERVENTIONS:
Device: Treadmilll — Hemodynamic changes before and after treadmill use
  Other Names: Saturation device; Sphygmomanometer
Other: mask — mask
  Arms: Hemodynamic changes due to mask use

SUMMARY:
The use of masks is a necessity due to the current pandemic conditions. The aim of the study is to examine the effects of the use of masks during effort on dyspnea and fatigue with hemodynamic parameters.

DETAILED DESCRIPTION:
The use of masks is a necessity due to the current pandemic conditions.There are studies on many parameters such as the effect of mask use on saturation (sp02), heart rate (HR) and blood pressure (BP). To determine whether there is a change in the performance of individuals in the masked and unmasked exercise test during exertion due to the scarcity of masked and unmasked maximal exercise tests and the insufficient measurement of the degree of fatigue felt, and to determine whether there is a change in the performance of individuals with and without mask, and to determine the hemodynamic responses in the body together with dyspnea and felt fatigue. This study will be conducted in order to examine the effect on

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to work,
* To be healthy,
* 18-25 age range.

Exclusion Criteria:

* Unstabil angina pectoris,
* Atrial arrhythmia,
* Uncontrollable asthma,
* Pa02 < 50 mmHg,
* PaCO2> 70mmHg,
* Individuals with valve disease
* Tachycardia, bradycardia,
* Individuals with a resting systolic blood pressure of 200 mmHg
* Smoking,
* Presence of effective clinical conditions such as nasal deviation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Measurement of blood pressure changes due to mask use | The period in which each participant is evaluated by taking the outcome criterion is 30-60 minutes.
  Blood pressure reading with sphygmomanometer.
Evaluation of dyspnea score | The period in which each participant is evaluated by taking the outcome criterion is 30-60 minutes.
  Dyspnea score was evaluated with the Modified Borg Scale. The Modified Borg Scale is a 0 to 10 numerical score used to measure dyspnea. 0 indicates minimum dyspnea and 10 indicates maximum dyspnea.
Evaluation of the degree of perceived fatigue | The period in which each participant is evaluated by taking the outcome criterion is 30-60 minutes.
  The degree of perceived fatigue was evaluated with the Modified Borg Scale. The Modified Borg Scale was used to assess perceived difficulty. The Modified Borg Scale is a numerical score from 0 to 10. 0 means minimum difficulty and 10 means maximum difficulty.
Measurement of oxygen saturation and heart rate changes due to mask use | The period in which each participant is evaluated by taking the outcome criterion is 30-60 minutes.
  Oxygen saturation and heart rate were recorded with a pulseoximetry device.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Karabıyık, Principal Investigator — Saglik Bilimleri Universitesi; Ayşegül Tunç, Principal Investigator — Saglik Bilimleri Universitesi; Zeynep Tanrıverdi, Principal Investigator — Saglik Bilimleri Universitesi; Selen Öztürk, Principal Investigator — Saglik Bilimleri Universitesi; Fulya Senem Karaahmetoğlu, Principal Investigator — Saglik Bilimleri Universitesi; Halit Çınarka, Principal Investigator — Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No